CLINICAL TRIAL: NCT07026396
Title: Creative Touch in Menstrual Attitude and Hygiene Behavior: A Drama Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esra Sayar, Dr, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-SBF-ES
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Creative Drama; Genital Hygiene; Menstrual Cycle; Adolescent
Keywords: adolescent; menstruation; creative drama

STUDY DESIGN:
Intervention Model Description: Randomize-control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): There will be no intervention in this group.
- Creative drama group (Experimental): In the intervention phase of the study, creative drama training was given to adolescents one day a week for 4 weeks. Before the training, permission was obtained from the families of the individuals, and only voluntary adolescents were allowed to participate. The empty classroom in the school was made suitable for creative drama activities. Adolescents gathered in the empty classroom one day a week, and the models and activity materials prepared by the researcher were taken to the classroom during the implementation week.
  Interventions: Other: Creative drama group

INTERVENTIONS:
Other: Creative drama group — In the intervention phase of the study, creative drama training was given to adolescents one day a week for 4 weeks. Before the training, permission was obtained from the families of the individuals, and only voluntary adolescents were allowed to participate. The empty classroom in the school was made suitable for creative drama activities. Adolescents gathered in the empty classroom one day a week, and the models and activity materials prepared by the researcher were taken to the classroom during the implementation week.
  Arms: Creative drama group

SUMMARY:
In this study, the effect of creative drama-based education on menstruation attitudes and genital hygiene behaviors of adolescent girls aged 10-14 years was investigated. After screening, a total of 64 students were included in the study. Data were collected using Personal Information Form, Genital Hygiene Behavior Scale and Menstruation Attitude Scale.The creative drama method can create an open and safe communication environment by reducing the embarrassment or shyness of young people when dealing with taboo subjects such as menstruation. This approach supported the perception of menstruation as a natural biological process and contributed to the participants developing a more positive attitude towards the subject.

DETAILED DESCRIPTION:
This study aimed to determine the effect of training with creative drama techniques on menstruation attitudes and genital hygiene behaviors of adolescent girls aged 10-14 years. Since the study will have one experimental and one control group, it was planned to have 40 students in each group. Eight students who did not attend 75% of the 4-week training and did not participate in the posttest were excluded from the experimental group, and eight students were excluded from the control group because they gave incomplete answers. A consort flow diagram was applied in the study. Personal Information Form, Genital Hygiene Behavior Scale (GHD-S), and Menstruation Attitude Scale (MAS) were used for data collection.

The creative drama method can create an open and safe communication environment by reducing the embarrassment or shyness of young people when dealing with taboo subjects such as menstruation. This approach supported the perception of menstruation as a natural biological process and contributed to the participants developing a more positive attitude towards the subject. Acquiring the right knowledge and attitudes about the menstrual period is critical for individuals to protect and improve their general health. It is known that effective health education is indispensable to meet the needs of this age group in solving problems specific to adolescence. Especially in the pubertal period, the vaginal epithelium of girls is thin and poor in glycogen due to low endogenous estrogen levels.This makes vaginal bacterial infections more common in this age group. Improper hygiene practices, such as the use of soap or shower gel for vaginal cleansing, systemic diseases such as diabetes, and the preference for tight, airtight underwear are among the factors that increase the risk of vaginal infections.For these reasons, providing adolescent girls with adequate knowledge about menstruation and genital hygiene should be an integral part of health education. Such education during adolescence helps young people develop healthy habits and is an important step towards preventing health problems they may face in the future.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 years old,
* Female gender
* No communication problems,
* Not having any cognitive, affective, or psychomotor disorders
* Voluntary participation in the study
* Exclusion Criteria
* Boys were not included in the study.
* The study did not include those who did not meet the inclusion criteria.

Exclusion Criteria:

* Boys were not included in the study.
* The study did not include those who did not meet the inclusion criteria.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — adolescent girls
Enrollment: 64 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Genital Hygiene Behavior Scale (GHD-S) | 5-10 minutes
  Genital Hygiene Behavior Scale (GHD-S): The scale, which has 23 items and three sub-dimensions, was developed by Karahan. The scale score range is 23-115, and as the scores increase, the correct genital hygiene behaviors increase. The Cronbach alpha value of the scale was determined as 0.80

SECONDARY OUTCOMES:
Menstruation Attitude Scale (MTS) | 5-10 minutes
  Menstruation Attitude Scale (MTS): The Turkish validity and reliability of the scale, which has 33 items and five sub-dimensions, was conducted by Kulakaç et al. The scale is Likert-type (1-7 points). As the score increases on the scale, menstrual behaviors increase. The scale Cronbach alpha value was determined as 0.70.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk university faculty of health sciences, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, we don't plan to share individual participant data

REFERENCES:
- [Background] Sayar SE, Capik C. The Effect of Health Belief Model-Based Creative Drama Education on Health Locus of Control and Smoking Perception in Adolescents: A Randomized Controlled Trial. Public Health Nurs. 2025 May-Jun;42(3):1343-1353. doi: 10.1111/phn.13550. Epub 2025 Mar 6. PMID 40047297
- [Background] Soleymani MR, Hemmati S, Ashrafi-Rizi H, Shahrzadi L. Comparison of the effects of storytelling and creative drama methods on children's awareness about personal hygiene. J Educ Health Promot. 2017 Oct 4;6:82. doi: 10.4103/jehp.jehp_56_16. eCollection 2017. PMID 29114550
- [Derived] Uzunlu S, Sayar SE, Calim GA, Capik C. Effect of a creative drama-based educational intervention on menstrual attitudes and genital hygiene behaviors in adolescent girls: a randomized controlled trial. BMC Public Health. 2026 Jan 20. doi: 10.1186/s12889-026-26331-6. Online ahead of print. PMID 41555265